CLINICAL TRIAL: NCT06167226
Title: Prediction of Ayurveda Prakriti and Vikriti Using Automatic Questionnaire and Digital Sensors
Brief Title: Understanding Ayurveda Disease Conditions and Treatment Responses
Status: Completed | Type: Observational
Sponsor: Ayurai Private Limited (Industry)
Collaborators: SRM Medical College Hospital & Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTRI/2021/12/038909
Record Dates: First submitted 2023-11-18; First posted 2023-12-12 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Type2diabetes; Rheumatoid Arthritis; Osteo Arthritis Knee; Skin Diseases; Gastric Ulcer; Neurodegenerative Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Skin Diseases; Stomach Ulcer; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Personalized Ayurveda treatment protocol — The treating physician decided and advised personalized Ayurveda treatment protocol based on disease and patient's condition
  Other Names: No other intervention name

SUMMARY:
The goal of this observational study is to assess Prakriti & Vikriti in patients visiting OPD of IIISM department, SRM hospital.

The main question[s] it aims to answer are:

* To evaluate Prakriti & Vikriti of patients using Prakriti & Vikriti questionnaire and with digital devices
* To correlate the determined Prakriti and Vikriti with the doctor's assessment along with clinical and biochemical parameters Participants will be advised to follow the treating physician's advice on medicines

DETAILED DESCRIPTION:
The Ayurveda is an ancient documented medical system originated in India. The Ayurveda stratified humans into 7 broad categories based on the phenotype features viz. Vata, Pitta, Kapha, Vatapitta, Vatakapha, Kaphapitta and Vatapittakapha Prakriti types. Also, the features of the disease conditions are clearly described based on the predominance of Vata, Pitta and Kapha or its combinations. Presently, the identification of Prakriti type and Vikriti status are basically subjective assessment. This study proposes to integrate the subjective assessment with objective digital signal parameters. This digital signatures would be useful in ML / AI based assessment and prediction of Prakriti type and Vikriti status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of various diseases visiting the OPD

Exclusion Criteria:

* Pregnancy and lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of various diseases visiting the OPD
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Complete blood count at 12 week | 12 weeks
  complete blood count, which includes red blood cell count, neutrophil count, eosinophil count, basophil count, lymphocyte count, monocyte count, and platelet count is a standard investigation to measure the abnormality in blood cells
Serum Urea | 12 weeks
  Measures urea, which is a investigation to measure the abnormality in kidney function
Serum creatinine | 12 weeks
  Measures creatinine, which is a investigation to measure the abnormality in kidney function
Lipid Profile | 12 weeks
  Lipid profile test includes Total cholesterol, LDL, HDL, Triglycerides, and non-HDL is a investigation to measure the abnormality in lipids
Cytokines (TNF- alpha, IFN-gamma, IL-1, IL-4, IL-6, IL-10) | 12 weeks
  Cytokines are inflammatory markers, measured to identify treatment effect in inflammation

SECONDARY OUTCOMES:
Pulse Plethysmography signals (PPG) - Finger PPG sensor | 12 weeks
  PPG is measured to identify pulse wave form changes before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: RC Sathish kumar, Principal Investigator — SRM Medical College Hospital & Research Centre
Locations (1):
- SRM Medical College Hospital & Research Centre, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identiﬁcation (text, tables, ﬁgures, and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publishing and for 3 years
Access Criteria: Researchers whose proposed use of the data has been approved by an independent review committee identiﬁed for this purpose.